CLINICAL TRIAL: NCT06576583
Title: Randomized, Controlled, Multi-center Phase II Clinical Trial for the Treatment of Patellofemoral Osteoarthritis With Nasal Chondrocyte-based Tissue Engineered Cartilage Implantation vs Current Standard of Care
Brief Title: Implantation of Engineered Cartilage Grafts for Treatment of Patellofemoral Osteoarthritis Versus Surgical Comparators.
Acronym: ENCANTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other); Wuerzburg University Hospital (Other); Medical University of Vienna (Other); Videoreha (Unknown); University of Oulu (Other); Theracell Laboratories (Unknown); Promove-Biotec GmbH (Unknown); Maastricht University (Other); Foundation National Reumafonds (Unknown); Angry@Arthritis (Unknown); University of Miami (Other); Geistlich Pharma AG (Industry); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-513683-25-00
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: Nasal chondrocytes; Tissue engineering; Knee cartilage; Patellofemoral osteoarthritis; Autologous Matrix Induced Chondrogenesis (AMIC); Patellofemoral arthroplasty (PFA)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Engineered cartilage graft (N-TEC)-Iwano grade 1-2 (Experimental): N-TEC is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membranes for 2 weeks to allow cells to produce extracellular matrix containing cartilage specific proteins. The IMP is implanted in the knee at the patellofemoral joint.
  Interventions: Biological: Engineered cartilage graft (N-TEC)
- Autologous Matrix Induced Chondrogenesis-Iwano grade 1-2 (Active Comparator): AMIC® Chondro-Gide® combines microfracturing (MFx) with the use of Chondro-Gide®, which covers and protects both the super clot resulting from MFx and the repair tissue.
  Interventions: Procedure: Autologous Matrix Induced Chondrogenesis (AMIC)
- Engineered cartilage graft (N-TEC)-Iwano grade 3-4 (Experimental): N-TEC is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membranes for 2 weeks to allow cells to produce extracellular matrix containing cartilage specific proteins. The IMP is implanted in the knee at the patellofemoral joint.
  Interventions: Biological: Engineered cartilage graft (N-TEC)
- Patellofemoral Arthroplasty (PFA)-Iwano grade 3-4 (Active Comparator): Patellofemoral Joint Prosthesis
  Interventions: Procedure: Patellofemoral Arthroplasty (PFA)

INTERVENTIONS:
Biological: Engineered cartilage graft (N-TEC) — Nasal chondrocytes based tissue engineered cartilage
  Arms: Engineered cartilage graft (N-TEC)-Iwano grade 1-2; Engineered cartilage graft (N-TEC)-Iwano grade 3-4
Procedure: Autologous Matrix Induced Chondrogenesis (AMIC) — Autologous Matrix Induced Chondrogenesis is performed through bone drilling and covering with Chondro-Gide® to attract bone marrow stem cells
  Arms: Autologous Matrix Induced Chondrogenesis-Iwano grade 1-2
Procedure: Patellofemoral Arthroplasty (PFA) — Surgical implantation of a medical device, Zimmer Gender Solutions Patellofemoral Joint Prosthesis.
  Arms: Patellofemoral Arthroplasty (PFA)-Iwano grade 3-4

SUMMARY:
ENCANTO is a randomized, controlled, multi-center phase II clinical trial for the treatment of patellofemoral osteoarthritis (PFOA) with an Advanced Therapy Medicinal Product (ATMP), nasal chondrocyte-based tissue engineered cartilage (N-TEC) implantation in comparison with current standard of care depending on the stage of osteoarthritis. The goal of this phase II trial is to evaluate the efficacy of N-TEC treatment in comparison to an active comparator Autologous Matrix Induced Chondrogenesis (AMIC) for early stage PFOA or patellofemoral arthroplasty (PFA) for late stage PFOA.

The N-TEC engineered cartilage graft is obtained by culturing expanded autologous nasal chondrocytes within a collagen type I/III membrane.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the most common causes for pain and disability with over 260 million people affected worldwide. Recent studies found that knee OA often starts in the patello-femoral compartment of the knee (PFOA) and is diagnosed in ~39% of people with knee pain aged above 30 years. Thus, PFOA and progression to full OA plays a crucial role in the reduction of quality of life of many people and in the raise of healthcare costs.

The goal of this multi-center phase II trial is to (i) evaluate the efficacy of N-TEC treatment in comparison to an active comparator Autologous Matrix Induced Chondrogenesis (AMIC) for early stage PFOA or patellofemoral arthroplasty (PFA) for late stage PFOA based on patient self-assessed questionnaires (Knee Injury and Osteoarthritis Outcome Score, KOOS) and (ii) verify the postulated mode of action, which is expected to be of regenerative nature and will be assessed by evaluation of disease-modification by x- ray and structural regeneration of the osteoarthritic joint destruction by MRI analysis. A total of 150 patients with early stage of PFOA (Iwano grade 1-2; 75 patients) or late stage of PFOA (Iwano grade 3-4; 75 patients) will be enrolled in 11 clinical centers and randomized to either N-TEC implantation or active comparator (AMIC or PFA).

ELIGIBILITY:
Inclusion Criteria:

* Patient age is ≥18 and ≤ 70 years at time of screening.
* Symptomatic PFOA grade 1-4 according to Iwano Classification
* Chondropathy Grade 3-4 according to ICRS classification of the patella, trochlea femoris or both
* Baseline score of <75 on the KOOS-5 subjective knee evaluation.
* Free range of motion of the affected knee joint or ≤ 5° of extension loss and minimum 125° flexion.
* Patient is willing and able to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments and to complete postoperative rehabilitation regimen.
* Minimum values for women: Haemoglobin 120g/l, Platelets 150G/l, INR<1.3
* Minimum values for men: Haemoglobin 140g/l, Platelets 150G/l, INR<1.3
* Patients have failed to demonstrate adequate response to non-pharmacological interventions (e.g. structured land-based exercise programs) and pharmacological first-line treatment such as topical NSAIDs

Exclusion Criteria:

* Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol or in a dependency or employment with the sponsor.
* Patient is unwilling, unable or lacking the capacity to provide informed consent
* Patient is unable to undergo magnetic resonance imaging (MRI)
* Prior surgical treatment of the target knee within 12 months (Note: prior diagnostic arthroscopy with debridement and lavage are acceptable within 12 months).
* Radiologically apparent degenerative joint disease of the tibiofemoral joint as determined by X-ray (Kellgren and Lawrence grade > 2) or MRI or pain in the tibiofemoral joint as assessed by clinical examination
* Patient has excessive varus or valgus deformity (>5°), unless corrected during implantation
* Patient has a symptomatic meniscus lesion (or removal exceeding ½), as indicated by clinical examination (joint line tenderness and McMurray test positive) and MRI.
* Patient has a body mass index (BMI) >35 kg/m2.
* Patient has chronic rheumatoid arthritis, and/or infectious arthritis
* Any concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee.
* Patient has a known immunological suppressive disorder or is taking systemic immunosuppressives.
* Patient had any intra-articular injections into the affected knee within the last 3 months before baseline visit
* Instability of anterior, posterior and/or collateral ligaments
* The patient has a HIV/AIDS infection. (regulatory requirement)
* The patient has an acute Treponema pallidum (syphilis) infection. (regulatory requirement)
* The patient has an active hepatitis B or C infection with verified antigens. Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded. (regulatory requirement)
* Patient is pregnant, breast feeding or anticipates becoming pregnant within 24 months after surgery.
* Patient is currently participating or has participated in any other clinical study within 3 months prior to the screening visit.
* Patient has known current or recent history of illicit drug or alcohol abuse or dependence defined as the continued use of alcohol or drugs despite the development of social, legal or health problems.
* Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.
* Known allergies for porcine collagen (scaffold), penicillin or streptomycin (manufacturing)
* Nail-patella syndrome
* Patients who will likely benefit from conservative therapy, such as physiotherapy, medical training therapy and pain medication
* Patients with increased anesthesiological and surgical risks (e.g. known or predicted difficult airway, myocardial infarction <60 days prior to surgery)
* Patients with increased bleeding risk (e.g. coagulopathies)
* Patients on anticoagulants whose anticoagulant therapy cannot be interrupted as appropriate to the given agent(s) and underlying condition
* Patients with any active infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS)-5 | 24 months
  Difference in 2-year change (baseline to 24 month follow-up) in the KOOS -5 score between patients undergoing N-TEC tissue implantation and patients receiving AMIC or PFA. Minimum score: 0 Maximum score: 100 (higher score means no knee problems)

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome questionnaire | until 24 months
  patient self reported questionnaire for pain
Knee Injury and Osteoarthritis Outcome questionnaire | Until 24 months
  patient self reported questionnaire for symptoms, activity of daily life, sports and quality of life Minimum score: 0 Maximum score: 100 (higher score means no knee problems)
Kujala questionnaire | Until 24 months
  patient self reported questionnaire for Anterior Knee Pain scale. Minimum score: 0 Maximum score: 100 (no knee problems)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Until 24 months
  Self reported questionnaire to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The instrument contains 24 items measuring 3 sub-scales: physical function (17 items), pain (5 items), and stiffness (2 items). Minimum score: 0 (no knee problems) Maximum score: 96 (worst knee problems)
EQ-5D-5L questionnaire | Until 24 months
  Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Global Rating Of Change (GROC) likert scale | Until 24 months
  Widely used score to assess whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change. Minimum score: -5 ; maximal score: +5.
Marx Activity Rating Scale (MARS) score | Until 24 months
  This activity-related patient-reported outcome measure is widely used to assess the activity of a patient after treatments of the knee. It assesses how often the patient performs activities (running, cutting, deceleration and pivoting) in his healthiest and more active state. Minimum score: 0; maximum score: 16.
Morphological analysis | Until 24 months
  Morphological analysis with assessment of whole cartilage volume (in mm3) by radiological assessment (MRI)
Collagen network organization | Until 24 months
  Collagen network organization with T2 mapping and RADIOMICS GLCM by radiological assessment (MRI)
Osteoarthritis grading | Until 24 months
  Osteoarthritis grade according to Iwano and Kellgren/Lawrence classification by radiological assessment (X-ray)
Biovigilance | Until 24 months
  Number of adverse events, adverse reactions based on severity, expectedness and relationship to treatment.

CONTACTS AND LOCATIONS:
Locations (11):
- Orthopedic Hospital Vienna-Speising, Vienna, Austria
- University Hospital Sveti Duh, Zagreb, Croatia
- Germany (2):
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Orthopedic Clinic König-Ludwig-Haus, Würzburg
- Italy (2):
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
- Maastricht University Medical Center, Maastricht, Netherlands
- Zeromski hospital, Krakow, Poland
- Department of Orthopaedics, University of Gothenburg (UGOT), Mölndal, Sweden
- Switzerland (2):
  - University Hospital Basel, Basel
  - Crossklinik, Basel

IPD SHARING:
Plan to Share IPD: No